CLINICAL TRIAL: NCT01704768
Title: COPE/Healthy Lifestyles for Teens: A School-Based RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01NR012171 (NIH); 1R01NR012171-01A2 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Lifestyle Behaviors; Depressive/Anxiety Symptoms
Keywords: Randomized Controlled Trial; School-Based Intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPE/Healthy Lifestyles TEEN Program (Experimental): COPE is a manualized 15-session educational and cognitive-behavioral skills building program guided by Cognitive Behavioral Theory with physical activity as a component of each session.
  Interventions: Behavioral: COPE/Healthy Lifestyles TEEN Program.
- Healthy Teens Attention Control Program (Placebo Comparator): Healthy Teens is an attention control program that controls for the time spent with the adolescents in the COPE group is essential to determining the efficacy of the experimental program.
  Interventions: Behavioral: Healthy Teens Attention Control Program

INTERVENTIONS:
Behavioral: COPE/Healthy Lifestyles TEEN Program. — The COPE Program is the intervention curriculum delivered to one arm of the study. Each session of COPE contains 15 to 20 minutes of physical activity (e.g., walking, dancing), not as an exercise training program, but rather to build beliefs/confidence in the teens that they can engage in and sustain some level of physical activity on a regular basis. Those healthy lifestyle intervention programs that have employed exercise interventions only have not led to sustained changes in healthy lifestyle behaviors. Our program is designed to enhance healthy lifestyle behaviors and sustain them because life-long cognitive-behavioral skills are taught in the program. Because the COPE TEEN program is completely manualized for the teens and instructors, it can be easily implemented by health teachers in high school settings.
  Other Names: Cognitive-Behavioral Skills Building
  Arms: COPE/Healthy Lifestyles TEEN Program
Behavioral: Healthy Teens Attention Control Program — The Healthy Teens program is an attention control program that will assist in ruling out alternative explanations of the mechanism by which the intervention works. It will be standardized like the COPE program to insure that it can be evaluated. It will be administered in a format like that of the COPE intervention program, and will include the same number and length of sessions, except for that it will not include the theoretical active components of CBT and will not include theoretical mechanisms to produce our hypothesized changes in outcomes. Teens in the attention control group also will receive the sessions in their required health class. The difference between the two programs will lie in the content of the sessions, with the Healthy Teens program being focused on safety and common health topics/issues for teens (e.g., road safety, skin care, acne, sun safety).
  Other Names: Educational
  Arms: Healthy Teens Attention Control Program

SUMMARY:
The prevention and treatment of obesity and mental health disorders in adolescence are two major public health problems in the United States today. To address the increasing incidence and adverse health outcomes associated with both obesity and mental health problems, a theory-based 15 session intervention program entitled COPE (Creating Opportunities for Personal Empowerment)/ Healthy Lifestyles TEEN(Thinking, Feeling, Emotions & Exercise), will be delivered within high school health classes in order to improve the physical and mental health outcomes of 800 culturally diverse adolescents (14 to 16 years of age).

DETAILED DESCRIPTION:
The prevention and treatment of obesity and mental health disorders in adolescence are two major public health problems in the United States (U.S.) today. The incidence of adolescents who are overweight or obese has increased dramatically over the past 20 years, with approximately 17.1 percent of teens now being overweight or obese. Furthermore, approximately 15 million children and adolescents (25 percent) in the U.S. have a mental health problem that is interfering with their functioning at home or at school, but less than 25 percent of those affected receive any treatment for these disorders. The prevalence rates of obesity and mental health problems are even higher in Hispanic teens, with studies suggesting that the two conditions often coexist in many youth. However, despite the rapidly increasing incidence of these two public health problems with their related health disparities and adverse health outcomes, there has been a paucity of theory based intervention studies conducted with adolescents in high schools to improve their healthy lifestyle behaviors as well as their physical and mental health outcomes. Unfortunately, physical and mental health services continue to be largely separated instead of integrated in the nation's healthcare system, which often leads to inadequate identification and treatment of these significant adolescent health problems.

Therefore, the goal of the proposed randomized controlled trial is to test the efficacy of the COPE(Creating Opportunities for Personal Empowerment)/Healthy Lifestyles TEEN (Thinking, Feeling, Emotions & Exercise) Program, an educational and cognitive-behavioral skills building intervention guided by cognitive behavior theory, on the healthy lifestyle behaviors and depressive symptoms of 800 culturally diverse adolescents enrolled in Phoenix, Arizona high schools. The specific aims of the study are to: (1) Use a randomized controlled trial to test the short- and more long-term efficacy of the COPE TEEN Program on key outcomes, including healthy lifestyles behaviors, depressive symptoms and body mass index percentage, (2) Examine the role of cognitive beliefs and perceived difficulty in leading a healthy lifestyle in mediating the effects of COPE on healthy lifestyle behaviors and depressive symptoms; and (3) Explore variables that may moderate the effects of the intervention on healthy lifestyle behaviors and depressive symptoms, including race/ethnicity, gender, SES, acculturation, and parental healthy lifestyle beliefs and behaviors. Six prior pilot studies support the need for this full scale clinical trial and the use of cognitive-behavioral skills building in promoting healthy lifestyles beliefs, behaviors and optimal mental health in teens.

ELIGIBILITY:
Inclusion Criteria:

* Teens and parents of any gender, ethnicity/race, or socioeconomic status.
* Teens 14 to 16 years of age who are freshmen and sophomores taking a health class at one of the participating high schools.
* Teens who assent to participation.
* Teens with a custodial parent who consents for themselves and their teen's participation in the study.
* Teens who can speak and read in English (educational instruction in Arizona High Schools is conducted in English)

Exclusion Criteria:

* Teens who are under age 14 will be excluded because:

  * They are not likely to be enrolled in high school, and
  * They are unlikely to have sufficient cognitive development to benefit from the proposed intervention
* Teens who are over age 16 will be excluded for two key reasons:

  * We believe that the cognitive development of and social expectations for older teens requires a more complex and flexible intervention than that proposed, and
  * Teens need to be available for 12 month follow-up sessions (our pilot studies indicated that this becomes less likely once teens are old enough to leave/graduate from high school, emancipate from parents, and/or leave home).

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1219 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index Percentage (BMI%) | Change from Baseline to 12-Month Post intervention
  Information regarding the participants age, gender, weight and height at time of data collection provide information to track BMI overtime.
Change in Healthy Lifestyle Behaviors | Change from Baseline to 12-Month Post intervention
  Healthy lifestyle behaviors will be measured with the Healthy Lifestyle Behaviors Scale developed for use in our preliminary studies. we also will employ pedometers to objectively quantify activity. Teens will be trained in the use of the pedometer. Pedometers provide a valid and reliable means to measure habitual physical activity in youth to be used as a measure of the students Healthy Lifestyles Behaviors.
Change in Depression and Anxiety Symptoms | Change from Baseline to 15-Week Post intervention
  Depression and Anxiety is measured utilizing the Beck Youth Inventory (2nd edition; BYI-II). This 100-item instrument for youth 7 to 18 years of age is a commercial product widely used in research and clinical settings that has well-established reliability, validity, and age, gender, and diagnostic-adjusted norms. It measures five constructs: (a) depressive symptoms, (b) anxiety symptoms, (c) anger, (d) disruptive behavior, and (e) self-concept.
Social Skills | 15-Week Post
  Social Skills are measured utilizing the Social Skills Rating System (SSRS), a commercial tool that is commonly utilized in research. The SSRS is completed by the student's health teacher.
Academic Performance | 15-Week Post
  Academic performance is measured utilizing the student's health class grades
Change in Body Mass Index Percentile (%) | Change from Baseline to 6-Month post intervention
  Information regarding the participants age, gender, weight and height at time of data collection provide information to track BMI overtime.
Change in Healthy Lifestyle Behaviors | Change from Baseline to 6-Month Post intervention
  Healthy lifestyle behaviors will be measured with the Healthy Lifestyle Behaviors Scale developed for use in our preliminary studies. we also will employ pedometers to objectively quantify activity. Teens will be trained in the use of the pedometer. Pedometers provide a valid and reliable means to measure habitual physical activity in youth to be used as a measure of the students Healthy Lifestyles Behaviors.
Change in Depression and Anxiety Symptoms | Change from Baseline to 6-Month Post intervention
  Depression and Anxiety is measured utilizing the Beck Youth Inventory (2nd edition; BYI-II). This 100-item instrument for youth 7 to 18 years of age is a commercial product widely used in research and clinical settings that has well-established reliability, validity, and age, gender, and diagnostic-adjusted norms. It measures five constructs: (a) depressive symptoms, (b) anxiety symptoms, (c) anger, (d) disruptive behavior, and (e) self-concept.
Change in Depression and Anxiety Symptoms | Change from Baseline to 12-Month Post intervention
  Depression and Anxiety is measured utilizing the Beck Youth Inventory (2nd edition; BYI-II). This 100-item instrument for youth 7 to 18 years of age is a commercial product widely used in research and clinical settings that has well-established reliability, validity, and age, gender, and diagnostic-adjusted norms. It measures five constructs: (a) depressive symptoms, (b) anxiety symptoms, (c) anger, (d) disruptive behavior, and (e) self-concept.

SECONDARY OUTCOMES:
Change in Healthy Lifestyles Beliefs | Change from Baseline to 15-Week Post intervention
  Healthy Lifestyles Beliefs are measured utilizing the Healthy Lifestyle Beliefs Scale (HLBS). The HLBS is a 16-item instrument that taps beliefs about various facets of maintaining a healthy lifestyle.
Change in Perceived Difficulty of Leading a Healthy Lifestyle | Change from Baseline to 15-Week Post intervention
  Perceived Difficulty is measured utilizing the Perceived Difficulty Scale. This instrument is a 12-item questionnaire that measures one's perceived difficulty in living a healthy lifestyle.
Change in Triglycerides (Lipid Panels) | Change from Baseline to 15-Week Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Triglycerides.
Change in Healthy Lifestyles Beliefs | Change from Baseline to 6-Months Post intervention
  Healthy Lifestyles Beliefs are measured utilizing the Healthy Lifestyle Beliefs Scale (HLBS). The HLBS is a 16-item instrument that taps beliefs about various facets of maintaining a healthy lifestyle.
Change in Healthy Lifestyles Beliefs | Change from Baseline to 12-Month Post intervention
  Healthy Lifestyles Beliefs are measured utilizing the Healthy Lifestyle Beliefs Scale (HLBS). The HLBS is a 16-item instrument that taps beliefs about various facets of maintaining a healthy lifestyle.
Change in Perceived Difficulty of Leading a Healthy Lifestyle | Change from Baseline to 6-Month Post intervention
  Perceived Difficulty is measured utilizing the Perceived Difficulty Scale. This instrument is a 12-item questionnaire that measures one's perceived difficulty in living a healthy lifestyle.
Change in Perceived Difficulty of Leading a Healthy Lifestyle | Change from Baseline to 12-Month Post intervention
  Perceived Difficulty is measured utilizing the Perceived Difficulty Scale. This instrument is a 12-item questionnaire that measures one's perceived difficulty in living a healthy lifestyle.
Change in Total Cholesterol (Lipid Panels) | Change from Baseline to 15-Week Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Total Cholesterol.
Change in High-Density Lipoprotein (HDL)(Lipid Panels) | Change from Baseline to 15-Week Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's High-Density Lipoprotein (HDL).
Change in Low-Density Lipoprotein (LDL) (Lipid Panels) | Change from Baseline to 15-Week Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Low-Density Lipoprotein (LDL).
Change in Triglycerides (Lipid Panels) | Change from Baseline to 6-Month Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Triglycerides.
Change in Total Cholesterol (Lipid Panels) | Change from Baseline to 6-Month Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Total Cholesterol.
Change in High-Density Lipoprotein (HDL) (Lipid Panels) | Change from Baseline to 6-Month Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's High-Density Lipoprotein (HDL).
Change in Low-Density Lipoprotein (LDL) (Lipid Panels) | Change from Baseline to 6-Month Post Intervention
  Participants whose BMI is at or above the 85th percentile are recruited to participate in the Lipid Panels. Participants who provide consent to participate in the Lipid Panels provide a blood sample through a finger stick which is tested for the participant's Low-Density Lipoprotein (LDL).

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette M Melnyk, PhD, RN, CPNP/PMHNP, FNAP FAAN, Principal Investigator — Ohio State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Melnyk BM, Kelly S, Tan A. Psychometric Properties of the Healthy Lifestyle Beliefs Scale for Adolescents. J Pediatr Health Care. 2021 May-Jun;35(3):285-291. doi: 10.1016/j.pedhc.2020.11.002. Epub 2021 Jan 29. PMID 33518442
- [Derived] McGovern CM, Militello LK, Arcoleo KJ, Melnyk BM. Factors Associated With Healthy Lifestyle Behaviors Among Adolescents. J Pediatr Health Care. 2018 Sep-Oct;32(5):473-480. doi: 10.1016/j.pedhc.2018.04.002. Epub 2018 Jun 22. PMID 29941235
- [Derived] Melnyk BM, Jacobson D, Kelly S, Belyea M, Shaibi G, Small L, O'Haver J, Marsiglia FF. Promoting healthy lifestyles in high school adolescents: a randomized controlled trial. Am J Prev Med. 2013 Oct;45(4):407-15. doi: 10.1016/j.amepre.2013.05.013. PMID 24050416